CLINICAL TRIAL: NCT02241928
Title: Role of Autologous Mononuclear Cell Therapy in Muscular Dystrophy
Brief Title: Stem Cell Therapy in Muscular Dystrophy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Neurogen Brain and Spine Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGBSI-14
Record Dates: First submitted 2014-09-12; First posted 2014-09-16 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Muscular Dystrophy
Keywords: Muscular Dystrophy; Autologous Mononuclear cell therapy; Stem Cell
MeSH Terms: conditions — Muscular Dystrophies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem Cell (Experimental): Bone marrow mononuclear cell transplantation
  Interventions: Biological: Stem Cell

INTERVENTIONS:
Biological: Stem Cell — Intrathecal Autologous bone marrow mononuclear cell transplantation

SUMMARY:
The purpose of this study was to analyze the effect of autologous bone marrow mononuclear cells in muscular dystrophy.

ELIGIBILITY:
Inclusion Criteria:

* age group of 6 months and above
* muscular dystrophy diagnosed on the basis of clinical presentation

Exclusion Criteria:

* presence of respiratory distress
* presence of acute infections such as Human Immunodeficient Virus/Hepatitis B Virus/Hepatitis C Virus
* malignancies
* acute medical conditions such as respiratory infection, fever, hemoglobin less than 8, bleeding tendency, bone marrow disorder, left ventricular ejection fraction < 30%
* pregnancy or breastfeeding

Ages: 6 Months to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Manual Muscle Testing | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Neurogen brain and spine institute, Navi Mumbai, Maharashtra, India